CLINICAL TRIAL: NCT01056146
Title: An Online Intervention for Families of Young Children With TBI: I-InTERACT
Brief Title: Interacting Together Everyday: Recovery After Childhood Traumatic Brain Injury (TBI) "I-InTERACT
Acronym: I-InTERACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H133G060167
Record Dates: First submitted 2010-01-20; First posted 2010-01-26 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-09

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; intracranial edema; brain edema; craniocerebral trauma; head injury; brain hemorrhage, traumatic; subdural hematoma; brain concussion; head injuries, closed; epidural hematoma; extra-axial hemorrhage; cortical contusion; Additional relevant MeSH terms:; Nervous System Diseases; Wounds and Injuries; Disorders of Environmental Origin; Central Nervous System Diseases; Trauma, Nervous System; Brain Diseases; Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema; Craniocerebral Trauma; Brain Hemorrhage, Traumatic; Hematoma, Subdural; Brain Concussion; Head Injuries, Closed; Hematoma, Epidural, Spinal; Brain Contusion; Nervous System Diseases; Wounds and Injuries; Disorders of Environmental Origin; Central Nervous System Diseases; Trauma, Nervous System; Brain Diseases; Brain Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet Resources Comparison (IRC) (Active Comparator): Participants will receive the Internet resource comparison group treatment
  Interventions: Behavioral: Internet Resources Comparison
- I-InTERACT (Experimental): Participants will receive the internet-based parenting skills program.
  Interventions: Behavioral: Internet-based Interacting Together Everyday: Recovery After Childhood TBI

INTERVENTIONS:
Behavioral: Internet-based Interacting Together Everyday: Recovery After Childhood TBI — Families in I-InTERACT will look through 10 web-sessions (like chapters) and participate in 10 family meetings focusing on education about traumatic brain injury, parenting skills, communication, behavior strategies, and stress management. Meetings will be conducted in their home using a computer hook-up with a trained therapist. Families will also be contacted two times per month by the counselor to discuss individual problems or concerns.
  Other Names: I-InTERACT
  Arms: I-InTERACT
Behavioral: Internet Resources Comparison — Families in the IRC group will receive computers, high speed internet access, and links to brain injury information and resources. The resources are available for families to access as often as they choose.
  Other Names: IRC
  Arms: Internet Resources Comparison (IRC)

SUMMARY:
The purpose of this study is to test an on-line intervention for families of young children who have experienced moderate or severe traumatic brain injury (TBI). Previous interventions were not designed to address the needs of young children with TBI, and feedback revealed a desire for more examples and materials appropriate for families of younger children. This project builds upon the investigators previous research by modifying the online intervention content to address the needs of young children with TBI. The goal of this project is to develop an intervention that will encourage positive parenting behaviors, improve child behaviors, and reduce parent distress and burden following TBI. The investigators hypothesize that the intervention group will exhibit more effective parenting skills as well as better child functioning and lower levels of parental distress at follow-up than will the active comparison group.

DETAILED DESCRIPTION:
Five million young children suffer from traumatic brain injury (TBI) each year resulting in new child behavior problems, parental distress, and family dysfunction. Recent studies provide evidence that online skill building interventions can reduce caregiver distress and improve child adjustment following TBI. The investigators hypothesize that the I-InTERACT group will exhibit more effective parenting skills as well as better child functioning and lower levels of parental distress at follow-up than will the IRC group. The investigators overarching goal is to reduce the risk of long-term behavioral problems and disability in young children following TBI by equipping parents with increased coping and parenting skills in a cost effective fashion. Findings will be disseminated via presentations and peer-reviewed publications, a website and newsletter, workshops with advocacy groups, and technical assistance to interested parties

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe TBI that occurred within the last 24 months
* Overnight hospital stay
* English-speaking
* Parent must be willing to provide informed consent

Exclusion Criteria:

* Child does not live with parents or guardian
* Child or parent has history of hospitalization for psychiatric problem
* Diagnosed with moderate or severe mental retardation, autism, or a significant developmental disability

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Parent Self Report Measures | 3 years
Videotaped parent-child interactions | 3 years

SECONDARY OUTCOMES:
Neuropsychological testing | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shari L. Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States